CLINICAL TRIAL: NCT02369900
Title: Esmolol to Treat the Hemodynamic Effects of Septic Shock
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding expired, low enrollments
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael N. Cocchi, MD, Michael N Cocchi MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000415; 15SDG22420010 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock; Hypotension; Tachycardia
Keywords: Esmolol; Septic Shock; Hypotension; Tachycardia
MeSH Terms: conditions — Shock, Septic; Hypotension; Tachycardia | interventions — esmolol; Adrenergic beta-Antagonists; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esmolol infusion (Active Comparator): Esmolol infusion for 24 hours. Esmolol will be titrated to a heart rate of 80 - 94 per minute, starting at 10mcg/kg/min and subsequently increasing every 20 minutes in increments of 10 mcg/kg/min (or slower at the discretion of the team) until target is achieved. The maximum allowed dose will be 300mcg/kg/min.
  Patients, irrespective of treatment group, will be managed at the discretion of the clinical team. BIDMC has internal guidelines for the management of septic shock which reflect the most recent 2012 Surviving Sepsis Campaign guidelines and are incorporated into the care of patients with septic shock in the ICUs
  Interventions: Drug: Esmolol
- Standard care, Saline (Placebo Comparator): Standard care (no esmolol). Patients, irrespective of treatment group, will be managed at the discretion of the clinical team. BIDMC has internal guidelines for the management of septic shock which reflect the most recent 2012 Surviving Sepsis Campaign guidelines and are incorporated into the care of patients with septic shock in the ICUs
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Esmolol
  Other Names: Beta Blocker
  Arms: Esmolol infusion
Other: Saline
  Other Names: Normal Saline
  Arms: Standard care, Saline

SUMMARY:
The main purpose of this study is to determine the effects of controlling the heart rate of patients with septic shock using an intravenous medication called esmolol.

DETAILED DESCRIPTION:
Septic shock is a leading cause of death around the world, with a mortality that often ranges 30-50% but in some locations may be even higher. Despite advances in critical care medicine over the last several decades, few therapeutic interventions have demonstrated mortality benefit in this population besides antimicrobial medications, intravenous fluids, and controlling the source of the infection; multiple agents which at one time showed promise have ultimately failed to deliver meaningful clinical benefit. As such, there is an ongoing need to identify therapeutic interventions which can modify the course of disease for these patients.

Septic shock is traditionally characterized by a hyperdynamic hemodynamic profile with a high cardiac output (CO) and low systemic vascular resistance (SVR) in association with excessive catecholamine stimulation. Tachycardia is a common finding in septic shock as an early compensatory mechanism to increase cardiac output in the setting of low SVR. Often tachycardia persists beyond the initial stages of septic shock, and has been associated with restricted diastolic ventricular filling, increased oxygen requirements, and tachycardia-induced cardiomyopathy, as well as myocardial depression, immunosuppression, and direct myocyte toxicity via calcium overload. Generally, clinical practice has been to avoid trying to control the tachycardic response for fear of worsening cardiac output and causing cardiovascular collapse. However, a recent single center randomized trial of the intravenous beta-1 adrenoreceptor antagonist esmolol demonstrated that control of heart rate to a more 'normal' range was safe, well-tolerated, and appeared beneficial, with a 30% reduction in mortality found in this trial.

While an intriguing concept with results that appear promising, further investigation among an ICU cohort in the United States is necessary before the administration of beta-blockade therapy to a patient in septic shock should be implemented in routine clinical practice. We hypothesize that the provision of esmolol to patients in vasopressor-dependent septic shock with tachycardia will lower the heart rate, thereby improving diastolic filling time and improving cardiac output, resulting in a reduction in need for vasopressor support. To test our hypothesis, we are conducting a Phase II randomized trial to determine if esmolol decreases vasopressor requirements (primary endpoint) and alters the inflammatory cascade as well as oxygen consumption in patients with septic shock (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Sepsis defined as suspected or confirmed infection with at least two systemic inflammatory response syndrome (SIRS) criteria
* Norepinephrine (minimum 0.1 mcg/kg/min) support to maintain a mean arterial pressure ≥ 65 mmHg despite appropriate volume resuscitation (as defined by the clinical team, however at least 30mL/kg intravenous fluid
* Heart rate ≥ 95 per minute for at least 2 hours prior to enrollment
* 6-24 hours since ICU admission

Exclusion Criteria:

* Intravenous β-blocker therapy prior to randomization
* Pronounced cardiac dysfunction (i.e. cardiac index [CI] ≤ 2.2 L/min/m2)
* Known significant valvular heart disease
* Research-protected populations (pregnant women, prisoners, intellectually disabled)
* Known "Do-not-resuscitate" or "do-not-intubate" order at the time of enrollment
* Infusion of epinephrine, dopamine, dobutamine or milrinone at time of enrollment
* Known allergy/sensitivity to esmolol or history of asthma/COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cocchi MN, Dargin J, Chase M, Patel PV, Grossestreuer A, Balaji L, Liu X, Moskowitz A, Berg K, Donnino MW. Esmolol to Treat the Hemodynamic Effects of Septic Shock: A Randomized Controlled Trial. Shock. 2022 Apr 1;57(4):508-517. doi: 10.1097/SHK.0000000000001905. PMID 35066509

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmolol Infusion: Esmolol infusion for 24 hours. Esmolol will be titrated to a heart rate of 80 - 94 per minute, starting at 10mcg/kg/min and subsequently increasing every 20 minutes in increments of 10 mcg/kg/min (or slower at the discretion of the team) until target is achieved. The maximum allowed dose will be 300mcg/kg/min.
  Patients, irrespective of treatment group, will be managed at the discretion of the clinical team. BIDMC has internal guidelines for the management of septic shock which reflect the most recent 2012 Surviving Sepsis Campaign guidelines and are incorporated into the care of patients with septic shock in the ICUs
  Esmolol
- Standard Care, Saline: Standard care (no esmolol). Patients, irrespective of treatment group, will be managed at the discretion of the clinical team. BIDMC has internal guidelines for the management of septic shock which reflect the most recent 2012 Surviving Sepsis Campaign guidelines and are incorporated into the care of patients with septic shock in the ICUs
  Saline
Period: Overall Study
Arm/Group | Esmolol Infusion | Standard Care, Saline
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmolol Infusion | Standard Care, Saline | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 14 | 24
  >=65 years | 8 | 8 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [59 to 71] | 62 [53 to 67] | 63 [58 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 18 | 31
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Need for Vasopressor Support, Measured as Mean Norepinephrine Equivalent Dose (mcg/kg/Min), at 6hr Time Point
Description: The primary endpoint will be mean norepinephrine equivalent dose (mcg/kg/min) at 6 hours after onset of study drug. For the vasopressor vasopressin, the dose of vasopressin was multiplied by 2.5 in order to create a norepinephrine equivalent dose. For the vasopressor phenylephrine, the dose of phenylephrine was divided by 10 in order to create a norepinephrine equivalent dose.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
mcg/kg/min | 0.30 (0.17) | 0.21 (0.19)

2. Secondary Outcome: Overall Need for Vasopressor Support
Description: While the primary endpoint will be mean norepinephrine dose at 6h, we will also measure mean vasopressor dose in groups at 12h and 24h.
Time Frame: 12 and 24 hours
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
mcg/kg/min
  12 hours | 0.31 (0.19) | 0.17 (0.17)
  24 hours | 0.24 (0.19) | 0.16 (0.17)

3. Secondary Outcome: Heart Rates Between Groups
Description: We will measure median heart rate at the 6 and 12h time points.
Time Frame: 6 and 12 hours
Measure: Median (Inter-Quartile Range); unit: beats per minutes
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
beats per minutes
  6 hours | 92 [89 to 104] | 98 [89 to 110]
  12 hours | 89 [79 to 105] | 96 [85 to 105]

4. Secondary Outcome: Time to Shock Reversal
Description: Time to shock reversal (cessation of all vasopressors for at least 12h).
Time Frame: Duration of hospitalization, limit 180 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
days | 3.9 [1.9 to 6.5] | 2.5 [1.5 to 6.1]

5. Secondary Outcome: Lactate
Description: Median percent change from baseline lactate measured at the 6, 12, and 24 hour time points after study initiation between groups. Percent change was calculated by subtracting the later lactate from the baseline lactate and dividing the difference by the baseline lactate (i.e. (baseline lactate - 6h lactate)/baseline lactate).
Time Frame: 6, 12, and 24 hours
Population: One patient in the standard care group was missing lactate levels at 6, 12, and 24 hours and one patient in the standard care group was missing a lactate level at 24 hours.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 21
percent change from baseline
  6 hours | 16.7 [2.7 to 22.2] | 0 [-21.4 to 19.3]
  12 hours | 27.5 [4.3 to 37.9] | 8.8 [-5.3 to 35.3]
  24 hours: number analyzed (Participants) | 18 | 20
  24 hours | 30.4 [12.1 to 50.0] | 19.1 [-18.2 to 37.1]

6. Secondary Outcome: Oxygen Consumption (VO2)
Description: To analyze the difference in oxygen consumption between groups at 12 hours, 24 hours and over time for patients who were on mechanical ventilation at enrollment, VO2 measurements were compared (standardized by bodyweight in kilograms) over time (recorded every minute from the time of study drug administration over a period of at least 24 hours) between groups using mixed linear model accounting for repeated measures. Using an unadjusted model, mean differences at 12 hours, 24 hours and for differences in the overall trend over time were tested.
Time Frame: 12 and 24 hours
Population: Only patients on mechanical ventilation who were able to be attached to the VO2 machine and had data within the first 24 hours were included.
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 6 | 9
mL/kg/min
  12 hours | 3.78 [3.09 to 4.21] | 4.29 [3.27 to 4.82]
  24 hours | 4.13 [2.74 to 6.32] | 4.83 [2.63 to 9.19]

7. Secondary Outcome: Interleukin-4
Description: To characterize effects of esmolol on inflammatory markers in patients with vasopressor-dependent septic shock, we compared log-transformed values of interleukin-4 at 12 and 24 hours and over time between groups using mixed linear model accounting for repeated measures and adjusting for pre-intervention levels.
Time Frame: 12 and 24 hours
Population: Blood was not able to be drawn from all patients at all time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
pg/mL
  12 hours: number analyzed (Participants) | 14 | 18
  12 hours | 0.027 [0.007 to 0.096] | 0.023 [0.018 to 0.069]
  24 hours: number analyzed (Participants) | 17 | 15
  24 hours | 0.016 [0.008 to 0.067] | 0.018 [0.011 to 0.086]

8. Secondary Outcome: Interleukin-6
Description: To characterize effects of esmolol on inflammatory markers in patients with vasopressor-dependent septic shock, we compared log-transformed values of interleukin-6 at 12 and 24 hours and over time between groups using mixed linear model accounting for repeated measures and adjusting for pre-intervention levels.
Time Frame: 12 and 24 hours
Population: Blood was not able to be drawn from all patients at all time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
pg/mL
  12 hours: number analyzed (Participants) | 16 | 20
  12 hours | 62.3 [22.5 to 190.5] | 78.3 [45.8 to 153.4]
  24 hours | 54.4 [18.1 to 242.4] | 39.0 [16.5 to 118.9]

9. Secondary Outcome: Interleukin-10
Description: To characterize effects of esmolol on inflammatory markers in patients with vasopressor-dependent septic shock, we compared log-transformed values of interleukin-10 at 12 and 24 hours and over time between groups using mixed linear model accounting for repeated measures and adjusting for pre-intervention levels.
Time Frame: 12 and 24 hours
Population: Blood was not able to be drawn from all patients at all time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
pg/mL
  12 hours: number analyzed (Participants) | 16 | 22
  12 hours | 3.5 [2.2 to 8.6] | 5.4 [1.9 to 13.0]
  24 hours | 3.4 [1.7 to 7.1] | 2.8 [1.4 to 6.0]

10. Secondary Outcome: TNF-alpha
Description: To characterize effects of esmolol on inflammatory markers in patients with vasopressor-dependent septic shock, we compared log-transformed values of TNF-alpha at 12 and 24 hours and over time between groups using mixed linear model accounting for repeated measures and adjusting for pre-intervention levels.
Time Frame: 12 and 24 hours
Population: Blood was not able to be drawn from all patients at all time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
pg/mL
  12 hours: number analyzed (Participants) | 16 | 20
  12 hours | 4.5 [2.3 to 8.9] | 8.7 [4.6 to 16.5]
  24 hours: number analyzed (Participants) | 18 | 18
  24 hours | 4.4 [2.8 to 6.9] | 7.5 [4.9 to 12.9]

11. Secondary Outcome: C-reactive Protein
Description: To characterize effects of esmolol on inflammatory markers in patients with vasopressor-dependent septic shock, we compared log-transformed values of C-reactive protein at 12 and 24 hours and over time between groups using mixed linear model accounting for repeated measures and adjusting for pre-intervention levels.
Time Frame: 12 and 24 hours
Population: Blood was not able to be drawn from all patients.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Esmolol Infusion | Standard Care, Saline
Number analyzed (Participants) | 18 | 22
pg/mL
  12 hours: number analyzed (Participants) | 16 | 20
  12 hours | 140.5 [101.8 to 191.8] | 170.2 [87.8 to 244.6]
  24 hours | 155.2 [74.0 to 201.8] | 189.7 [105.4 to 217.5]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Esmolol Infusion | Standard Care, Saline
All-Cause Mortality (participants affected / at risk) | 6/18 | 8/22
Serious Adverse Events (participants affected / at risk) | 4/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmolol Infusion (N=18) | Standard Care, Saline (N=22)
Decrease in Cardiac Index (Cardiac disorders) | 4 (4) | 0 (0) — During intervention, the patient's CI dropped below 2.1. The esmolol medication was stopped per protocol.
Abnormal Heart Rhythym (Cardiac disorders) | 1 (1) | 0 (0) — Patient had incidents of supraventricular tachycardia. The clinical team decided to continue esmolol treatment as the event was deemed unrelated to study protocol.
PEA arrest (General disorders) | 1 (1) | 0 (0) — An enrolled subject experienced a brief PEA arrest during turning. The arrest was attributed to a kinked endotracheal tube during turning and unrelated to study protocol.

LIMITATIONS AND CAVEATS:
The trial ended early due to slow enrollments and ending of funding before the target enrollment was reached. Many patients with septic shock were excluded because of the absence of tachycardia, or due to the presence of myocardial dysfunction. We did not collect echocardiographic data. Patients in the esmolol arm had differing exposures to esmolol, based on variable dosing and duration due to individual patient characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT02369900/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT02369900/SAP_001.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT02369900/ICF_002.pdf